CLINICAL TRIAL: NCT03011125
Title: A Phase 1 Double-blind, Dose-escalation, Placebo-controlled Tolerance Study in Healthy Chinese Adults After Single Intravenous Administration of Dexlansoprazole
Brief Title: A Clinical Trial to Evaluate the Safety and Tolerability of Dexlansoprazole Injection in Healthy Chinese Adults (Part 1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Jiangsu Aosaikang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASKC263-LC-1
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-01

CONDITIONS: Safety Issues
MeSH Terms: interventions — Dexlansoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Other: placebo
- Dexlansoprazole Injection (Experimental)
  Interventions: Drug: dexlansoprazole injection

INTERVENTIONS:
Drug: dexlansoprazole injection
  Arms: Dexlansoprazole Injection
Other: placebo
  Arms: placebo

SUMMARY:
This is a single center, randomized, double-blind, dose-escalation, placebo-controlled phase 1 clinical trial. This study will determine the safety and side-effect profile of an investigational dexlansoprazole injection after single intravenous administration in healthy Chinese adults.

DETAILED DESCRIPTION:
This is a single center, double-blind, dose-escalation, placebo-controlled clinical trial. Dose escalation will be proceeded according to 3+3 design in five predefined dosing groups. After completion of the 90mg dosing study, dose-escalation will be stopped, even though MTD is not be observed. A total of 28 participants is scheduled to be recruited. The whole follow-up period for each participant will be 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 Years;
* Male (weight ≥50kg) or female (weight ≥45kg);
* BMI between 19~28 kg/m2;
* Healthy subjects (at screening);
* Subject who totally understand the aim and progress of this clinical trial, make decision by his/her free will, and signed a consent form to follow the progress.

Exclusion Criteria:

* Allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator;
* Subject who has past or present history of any serious diseases, including (but not limited to) digestive, cardiovascular, respiratory, urinary, musculoskeletal, endocrine, psychiatric or neurological, hematologic, immunological or metabolic disorders;
* Medical examination, laboratory tests or ECG judged by the investigator to differ significantly from normal clinical values;
* HIV, HBV, or syphilis positive;
* Drug dependency or abuse;
* Heavy smokers (>5 cigarettes per day);
* Alcohol use;
* Participation in another study with an investigational drug within the last 3 months preceding this study;
* Blood donation within the last 2 months (>= 400 ml), or have a plan to donate blood within 1 month after this study;
* Intake of any other drug which might influence the results of the trial during two weeks previous to the start of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-03-09 (Actual); Study Completion 2017-03-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3 days
  Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lihua Wu, Doctor, Principal Investigator — First Affiliated Hospital of Zhejiang University

IPD SHARING:
Plan to Share IPD: No